CLINICAL TRIAL: NCT06577493
Title: Effectiveness of Phenazopyridine for Pain Following Urodynamics
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of South Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 007227
Record Dates: First submitted 2024-07-25; First posted 2024-08-29 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Pain After Urodynamic Testing
MeSH Terms: interventions — Phenazopyridine

STUDY DESIGN:
Intervention Model Description: Patients will be randomized into experimental or control groups
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Experimental Arm (Experimental): Patient to take two 99.5mg phenazopyridine hydrochloride (AZO) for a total of 199 mg by mouth once immediately prior to the start of urodynamic testing.
  Interventions: Drug: Phenazopyridine Hydrochloride 99.5 MG
- Control Arm (No Intervention): Patient to not receive any medication prior to the start of urodynamic testing.

INTERVENTIONS:
Drug: Phenazopyridine Hydrochloride 99.5 MG — Experimental arm to take two 99.5 mg phenazopyridine hydrochloride by mouth for a total of 199mg immediately prior to start of urodynamic testing
  Other Names: AZO
  Arms: Experimental Arm

SUMMARY:
The purpose of the study is to determine if taking phenazopyridine (AZO) at the time of urodynamic study testing will decrease pain experienced by patients after undergoing urodynamic testing.

ELIGIBILITY:
Inclusion Criteria:

* ability to provide informed consent
* ability to complete visual analog scale
* requiring urodynamic testing
* 18 years of age or older
* must be able to read and write in English or Spanish

Exclusion Criteria:

* allergy to phenazopyridine
* a urinary tract infection in the prior 2 weeks
* women who did not undergo urodynamic testing
* patient less than 18 years old
* patients with known (noted in patient chart and verbally asked) severe renal insufficiency with GFR <50 mL/min,
* patients with known (noted in patient chart and verbally asked) severe hepatitis
* patients with known (noted in patient chart and verbally asked) G6PD deficiency
* history of fibromyalgia
* history of interstitial cystitis
* non English or Spanish speaking

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2024-12-17 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Difference in pain scores, as measured by visual analog scale between study groups at 4 to 6 hours after urodynamic testing | 4 to 6 hours after testing
  Scores are measured on a 100mm VAS. The VAS ranges from 0 to 100 with 0 indicating no pain and higher scores indicating greater pain.

SECONDARY OUTCOMES:
Difference in anxiety scores, as measured by visual analog scale between study groups at predetermined time points. | baseline (immediately prior to testing), immediately after testing, 4 to 6 hours after testing
  Scores are measured on a 100mm VAS. The VAS ranges from 0 to 100 with 0 indicating no anxiety and higher scores indicating greater anxiety.
Difference in Urodynamic voiding parameters between experimental group and known normal values - UDS procedure length time | at time of testing
  Determine if preprocedural phenazopyridine has any change on normal urodynamic voiding parameters (UDS procedure length time) recorded in minutes
Difference in Urodynamic voiding parameters between experimental group and known normal values - first sensation | at time of testing
  Determine if preprocedural phenazopyridine has any change on normal urodynamic voiding parameters (first sensation) measured in mL
Difference in Urodynamic voiding parameters between experimental group and known normal values - first desire | at time of testing
  Determine if preprocedural phenazopyridine has any change on normal urodynamic voiding parameters (first desire) measured in mL
Difference in Urodynamic voiding parameters between experimental group and known normal values - strong desire | at time of testing
  Determine if preprocedural phenazopyridine has any change on normal urodynamic voiding parameters (strong desire) measured in mL
Difference in Urodynamic voiding parameters between experimental group and known normal values - capacity | at time of testing
  Determine if preprocedural phenazopyridine has any change on normal urodynamic voiding parameters (capacity) measured in mL
Difference in Urodynamic voiding parameters between experimental group and known normal values - valsalva leak point pressure | at time of testing
  Determine if preprocedural phenazopyridine has any change on normal urodynamic voiding parameters (valsalva leak point pressure) recorded in cmH20
Difference in Urodynamic voiding parameters between experimental group and known normal values - max flow rate | at time of testing
  Determine if preprocedural phenazopyridine has any change on normal urodynamic voiding parameters (max flow rate) is measured in mL/second
Difference in Urodynamic voiding parameters between experimental group and known normal values - voided volume | at time of testing
  Determine if preprocedural phenazopyridine has any change on normal urodynamic voiding parameters (voided volume) is measured in mL
Difference in Urodynamic voiding parameters between experimental group and known normal values - void time | at time of testing
  Determine if preprocedural phenazopyridine has any change on normal urodynamic voiding parameters (void time) is measured in minutes:seconds
Difference in Urodynamic voiding parameters between experimental group and known normal values - flow time | at time of testing
  Determine if preprocedural phenazopyridine has any change on normal urodynamic voiding parameters (flow time) is measured in minutes:seconds
Difference in Urodynamic voiding parameters between experimental group and known normal values - average flow rate | at time of testing
  Determine if preprocedural phenazopyridine has any change on normal urodynamic voiding parameters (average flow rate) is measured in mL/seconds
Difference in Urodynamic voiding parameters between experimental group and known normal values - time to max flow | at time of testing
  Determine if preprocedural phenazopyridine has any change on normal urodynamic voiding parameters (time to max flow) is measured in minutes:seconds
Difference in Urodynamic voiding parameters between experimental group and known normal values - max detrusor pressure | at time of testing
  Determine if preprocedural phenazopyridine has any change on normal urodynamic voiding parameters (max detrusor pressure) is measured in cm H20
Difference in Urodynamic voiding parameters between experimental group and known normal values - post void residual volume | at time of testing
  Determine if preprocedural phenazopyridine has any change on normal urodynamic voiding parameters (post void residual volume) is measured in mL
Number of patient communications | Per single participant (24 hours after completion of UDS testing)
  Count the number of patient communications after the completion of study
Would patients repeat urodynamic testing | 4 to 6 hours after testing
  Evaluate patients' willingness to undergo urodynamic testing again measured by a 1 to 5 likert scale with 1 being not at all likely and 5 being very likely

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth A Wilkinson, MD, Principal Investigator — University of South Florida
Locations (1):
- University of South Florida South Tampa Center, Tampa, Florida, United States

DOCUMENTS (1):
  • Informed Consent Form (2024-05-22): https://cdn.clinicaltrials.gov/large-docs/93/NCT06577493/ICF_000.pdf